CLINICAL TRIAL: NCT00005018
Title: A Phase IV 48-Week, Randomized, Open-Label, Multicenter Trial of Abacavir (300mg BID)/Efavirenz (600mg QD)/Didanosine (400mg QD) +/- Hydroxyurea (500mg BID) in HIV-1 Infected Subjects Failing Initial Therapy With 3TC/ZDV (or d4T) +/- Protease Inhibitor(s)
Brief Title: Safety and Effectiveness of a Combination Anti-HIV Drug Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 238R; NZTA4008
Record Dates: First submitted 2000-04-04; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: HIV Infections
Keywords: HIV-1; Didanosine; Drug Therapy, Combination; Zidovudine; Stavudine; HIV Protease Inhibitors; Hydroxyurea; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Hydroxyurea; abacavir; efavirenz; Didanosine

INTERVENTIONS:
Drug: Hydroxyurea
Drug: Abacavir sulfate
Drug: Efavirenz
Drug: Didanosine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give HIV-positive patients a combination of anti-HIV drugs (abacavir [ABC] plus efavirenz [EFV] plus didanosine [ddI]) with and without hydroxyurea (HU).

DETAILED DESCRIPTION:
Patients are randomized into one of two treatment arms: ABC/EFV/ddI or ABC/EFV/ddI/HU. In the second treatment arm, patients are further randomized to receive HU beginning at Baseline, when ABC/EFV/ddI is started, or at Week 8. Delaying HU may help offset the cytopenic effect of HU, as reflected in a blunted CD4 cell response. Patients are stratified according to their screening plasma HIV-1 RNA level (400 to 10,000 copies/ml and more than 10,000 to 100,000 copies/ml). Participants in the study receive study-related exams, lab tests, and study medications at no cost over the 48-week treatment period. The safety and effectiveness of the non-protease inhibitor rescue therapy is evaluated routinely by measuring viral load and the CD4 cell count, as well as the side effects caused by the medications. All of the medications are approved by the FDA and are not considered investigational.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are taking lamivudine (3TC) plus either zidovudine (ZDV) or stavudine (d4T). Patients may also be taking one or two protease inhibitors (PIs). (Patients will qualify if drug substitutions were made or if the drugs were stopped for up to 2 months under certain conditions.)
* Have a viral load of 400 copies/ml or more (treatment failure) after 16 weeks of this treatment.
* Have a viral load between 400 and 100,000 copies/ml.
* Have a CD4 cell count of 100 cells/mm3 or more.
* Have consent of a parent or guardian (if under 18).
* Agree to use a barrier form of birth control (such as condoms) during the study.
* Are at least 13 years old.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are unable to take medications by mouth.
* Have certain opportunistic (AIDS-related) infections or diseases.
* Have certain serious medical conditions such as diabetes or a disease of the liver, pancreas, or heart.
* Have a history of lymphoma.
* Have had peripheral neuropathy (a painful condition affecting the nervous system) within 2 months of study entry.
* Have been taking anti-HIV drugs for more than 1.5 years without an effect on HIV levels.
* Have ever taken ABC, ddI, or a type of anti-HIV drug called an NNRTI (such as EFV).
* Are unable to complete all 48 weeks of the study or take all of the study drugs.
* Are receiving certain other investigational treatments.
* Are receiving radiation therapy or chemotherapy within 8 weeks of study entry, or plan to receive one of these treatments during the study. (Local treatment for Kaposi's sarcoma is allowed.)
* Are taking certain medications including those that might affect the immune system or HIV levels.
* Have received a vaccine within 8 weeks of study entry or an HIV vaccine within 3 months of study entry.
* Are pregnant or breast-feeding.
* Abuse alcohol or drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1999-07; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - East Bay AIDS Ctr, Berkeley, California
  - Pacific Oaks Research, Beverly Hills, California
  - Altamed Medical Health Services, Los Angeles, California
  - St Lukes Medical Group, San Diego, California
  - Pacific Horizons Med Group, San Francisco, California
  - Gary Richmond MD, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Saint Josephs Comprehensive Research Institute, Tampa, Florida
  - Northstar Med Clinic, Chicago, Illinois
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - Boston Med Ctr / Evans - 556, Boston, Massachusetts
  - CRI of New England, Brookline, Massachusetts
  - Univ of Nebraska Medical Ctr, Omaha, Nebraska
  - Beth Israel Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Univ of North Carolina / Infectious Disease Division, Chapel Hill, North Carolina
  - Univ of NC Infectious Diseases, Wilmington, North Carolina
  - Anderson Clinical Research Inc, Reading, Pennsylvania
  - Miriam Hosp, Providence, Rhode Island
  - Burnside Clinic, Columbia, South Carolina
  - Univ of Texas Med Branch, Galveston, Texas
  - Univ of Texas / Thomas Street Clinic, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia